CLINICAL TRIAL: NCT05380440
Title: Preventing Parental Opioid and/or Methamphetamine Addiction Within DHS-Involved Families: PRE-FAIR
Acronym: PRE-FAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lisa Saldana, Senior Research Scientist, Chestnut Health Systems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1174-0623; 7UH3DA050193 (NIH)
Record Dates: First submitted 2021-07-12; First posted 2022-05-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Opioid-Related Disorders; Stimulant-Related Disorder; Child Neglect; Mental Health Impairment
Keywords: Substance-Related Disorders; Preventive Health Services; Opioid-Related Disorders; Amphetamine-Related Disorders; Child Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Amphetamine-Related Disorders | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRE-FAIR (Experimental): Participants in this arm will receive the PRE-FAIR intervention.
  Interventions: Behavioral: Prevention Adaptation of Families Actively Improving Relationships (PRE-FAIR)
- Control (Active Comparator): Participants in this arm will receive services standard case management and services .
  Interventions: Behavioral: Standard Case Management and Referral

INTERVENTIONS:
Behavioral: Prevention Adaptation of Families Actively Improving Relationships (PRE-FAIR) — FAIR is a behavioral intervention to treat parental substance use and child neglect for families involved in the child welfare system. This project will adapt the existing FAIR intervention for prevention (PRE-FAIR). FAIR involves four major treatment components, supported by ongoing purposeful engagement : (1) Substance use treatment including contingency management and positive reinforcement, frequent urinalysis, relationship building, day planning, healthy environments and peer choices, and refusal skills; (2) Mental health treatment including cognitive behavioral therapy, developing healthy coping skills, emotion regulation skills, exposure therapy, and referral for medication management; (3) Parent management training including parenting skills, nurturing and attachment, reinforcement, emotion regulation, supervision, structure, non-harsh discipline, and nutrition; and (4) Resource building and provision of ancillary supports including assistance with housing and employment.
  Arms: PRE-FAIR
Behavioral: Standard Case Management and Referral — Parents will be referred for a substance use and mental health assessment with possible resulting treatment. Child Welfare treatment plans typically include a series of recommendations, including parenting classes, securing safe housing, psychosocial treatment (e.g., domestic violence), accessing self-sufficiency services (e.g., food stamps, WIC), securing employment or education, and meeting court dates and requirements.
  Arms: Control

SUMMARY:
Young parents aged 16 to 30, involved in the DHS system for child welfare or self-sufficiency needs are at risk for opioid use disorder and/or methamphetamine use disorder (OUD; MUD). Those identified as engaging in opioid or methamphetamine misuse are at high risk for escalation. Children of parents with OUD and MUD are at-risk for entering into foster care. Oregon is one state particularly affected by this challenge. The proposed research offers one potential solution by adapting and evaluating a recently developed treatment for parental OUD and MUD, for prevention. This study seeks to collaborate with Oregon Department of Humans Services (DHS) leadership to deliver a new outpatient prevention program to high-risk, young, parents. The Prevention Adaptation of Families Actively Improving Relationships (PRE-FAIR) program will include community-based mental health, parent management, and ancillary needs treatment, and ongoing monitoring and prevention services for opioid and methamphetamine use. This study will randomize 240 parents, aged 16 to 30, to receive PRE-FAIR or standard case management and referral, in two counties in Oregon. Outcomes will include an evaluation of the effectiveness of PRE-FAIR in addressing risk factors associated with substance use disorders in DHS-involved populations, OUD and MUD outcomes, and implementation outcomes including implementation process and milestones, and program delivery outcomes. Intervention and Implementation costs will be assessed, and the benefit of PRE-FAIR will be evaluated in relation to standard services, but also in relation to capacity and population needs. Study hypotheses are: (1) Parents randomized to PRE-FAIR will be less likely to escalate opioid and/or methamphetamine use, and to receive a diagnosis of OUD and/or MUD; (2) Parents randomized to PRE-FAIR will experience significant reductions in mental health, parent skills, and ancillary needs compared to those receiving standard services; (3) Counties will follow the implementation plan developed in collaboration between study team members and state leadership, and that doing so will yield successful implementation of PRE-FAIR; and (4) Implementation and intervention costs for PRE-FAIR will demonstrate a benefit for offering PRE-FAIR compared to standard services, particularly in rural communities where capacity influences service delivery decisions.

DETAILED DESCRIPTION:
The Families Actively Improving Relationships (FAIR) program is a recently developed, rigorously evaluated, intensive outpatient treatment program for parents involved in the child welfare system for parental opioid and/or amphetamine type substance use disorder-methamphetamine (OUD; MUD). Outcomes from the FAIR effectiveness trial suggest the potential for FAIR to be adapted as a prevention program for parents involved with child welfare and self-sufficiency systems, and to be implemented in counties with low service availability and access. This exploratory-developmental phased project dedicates a year of activities toward collaborating with Oregon state Department of Human Services (DHS) partners and leadership to develop a plan for adaptation, recruitment, and implementation of FAIR for prevention (PRE-FAIR). The investigative team-with expertise in intervention development and clinical effectiveness trials, implementation science, decision science, health economics, and including DHS leadership-will work in collaboration with the Coordinating Center to develop strategies to identify, reach, and engage parents involved in the DHS system, aged 16 to 30, who are at-risk for escalation of misuse or development of OUD and/or MUD; and develop and adapt FAIR to prevent initiation of opioid and/or methamphetamine misuse and escalation to disorder. Following the completion of a set of concrete milestones during the first year, the project will conduct a Hybrid I randomized clinical trial, to evaluate the PRE-FAIR program and its implementation. Across two counties, parents referred by DHS for opioid or methamphetamine use or misuse with risk for escalation (n = 240), will be recruited and followed longitudinally for 24 months. Parents will be randomized to receive PRE-FAIR or standard case management and referral (STAND). Overarching goals of this study phase are to test the effectiveness of the adaptations designed in the previous phase and to build upon state collaborations-specifically, to: Evaluate the effectiveness of PRE-FAIR in preventing DHS-involved parents, aged 16 to 30, from initiating misuse or escalating opioid and/or methamphetamine use; Examine and assess the implementation of PRE-FAIR in the county-driven DHS system to inform sustainability plans; and Assess the implementation and intervention costs associated with the adoption of PRE-FAIR. Outcomes from this project will inform further refinement of protocols and the potential for broader scale-up of PRE-FAIR.

ELIGIBILITY:
Inclusion Criteria:

1. Risk for opioid or methamphetamine misuse or escalation of use
2. Parent of a child 0-18.
3. Involvement or risk for involvement with self-sufficiency or child welfare systems.
4. Aged 16 to 30 at date of intake assessment.
5. Enrolled in Oregon Health Plan
6. Child in home or reunification plan in place.
7. Lives in a participating Oregon county.

Exclusion Criteria:

* Used methamphetamines or opioids 4 or more times in past year
* Active diagnosis of a methamphetamine or opioid use disorder

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 241 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Change in opioid or methamphetamine use measured from Baseline to 24 months post-baseline | Baseline; 4-, 8-, 12-, 18-, and 24- months post Baseline
  Any opioid or methamphetamine use in the past 30 days measured by the Addiction Severity Index
Completion of Key Intervention Implementation Activities Over the Course of the Study | Duration of the study, up to 4 years
  Measure of implementation progress as measured by the Stages of Implementation Completion (SIC).
Costs Associated with Key Intervention Implementation Activities Over the Course of the Study | Duration of the study, up to 4 years
  Implementation costs associated with adoption of PRE-FAIR as measured by the Cost of Implementing New Strategies (COINS).
Mean changes in parent drug cravings and stress as measured by the Parent Daily Report | Baseline, monthly for 18-months post-Baseline, 24-months post-Baseline
  Parental stress and drug cravings as measured by the Parent Daily Report (PDR). Measured monthly from Baseline to 18-months post-Baseline and at 24-months post-Baseline.
Mean changes in behavioral health services utilization | up to 24- months
  Behavioral health services utilization (mental health, substance use) including visits assessed in the Service Utilization Survey and PRE-FAIR visits assessed in the coach portal software. Measured at Baseline, 4-, 8-, 12-, 18-, and 24-Months Post-Baseline.

SECONDARY OUTCOMES:
Mean Changes in Drug Use Frequency and Severity from Baseline to 24-months Post-Baseline | Baseline to 24-months Post-Baseline
  Drug use frequency and severity measured through the Addiction Severity Index's (ASI) Drug Use subscale. Measured at Baseline, 4-, 8-, 12-, 18-, and 24-Months Post-Baseline.
Changes in probability of opioid or methamphetamine use drug use as measured by Urinalysis testing | Baseline; 4-, 8-, 12-, 18-, and 24- months post Baseline
  Urinalysis based multi-drug panel using the ICUP Drug Screening device. Measured at Baseline, 4-, 8-, 12-, 18-, and 24-Months Post-Baseline.
Mean Changes From Baseline in Parenting Behaviors as Assessed by the BCAP at 24-months Post-Baseline | Baseline to 24-months Post-Baseline
  Parenting behaviors as measured by the Brief Child Abuse Potential Inventory (BCAP). Measured at Baseline, 4-, 8-, 12-, 18-, and 24-Months Post-Baseline.
Mean changes in anxiety symptoms reported as measured by the General Anxiety Disorder-7 (GAD-7) | Baseline; 4-, 8-, 12-, 18-, and 24- months post Baseline
  Anxiety symptoms as measured by the General Anxiety Disorder-7 (GAD-7). Measured at Baseline, 4-, 8-, 12-, 18-, and 24-Months Post-Baseline.
Mean changes in depression severity as measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline; 4-, 8-, 12-, 18-, and 24- months post Baseline
  Depression severity as measured by the Patient Health Questionnaire-9 (PHQ-9). Measured at Baseline, 4-, 8-, 12-, 18-, and 24-Months Post-Baseline.
Mean changes in post-traumatic stress and psychological effects of trauma as measured by the Trauma Symptom Inventory-2 (TSI-2) | Baseline; 4-, 8-, 12-, 18-, and 24- months post Baseline
  Measure of PTSD symptoms and psychological effects of trauma as measured by the Trauma Symptoms Inventory-2 (TSI-2). Measured at Baseline, 4-, 8-, 12-, 18-, and 24-Months Post-Baseline.
Mean Changes in Mental Health Symptoms from Baseline to 24-months Post-Baseline | Baseline to 24-months Post-Baseline
  Mental health symptoms as measured by the Brief Symptom Inventory (BSI). Sum of responses to 53 Likert-type items, range 0-24. Measured at Baseline, 4-, 8-, 12-, 18-, and 24-Months Post-Baseline.
Mean changes in parenting stress as measured by Parenting Stress Inventory | Baseline; 4-, 8-, 12-, 18-, and 24- months post Baseline
  Parenting stress as measured by the Parent Stress Inventory (PSI). Measured at Baseline, 4-, 8-, 12-, 18-, and 24-Months Post-Baseline.
Descriptive Measures of FAIR Program Delivery | Duration of the study, up to 4 years
  Descriptives of FAIR program delivery including: fidelity, attendance, caseload size, case characteristics, and session characteristics will be collected.
Mean Levels of Client Satisfaction with Services at the End of Treatment | End of treatment, average of 9 months
  Participants' self-reported perceptions of services as measured by the Client Satisfaction with Services Questionnaire (CSQ).

OTHER OUTCOMES:
Program Fidelity Ratings | Duration of study, up to 4 years
  Fidelity ratings of FAIR program fidelity as measured through behavioral coding of FAIR supervision sessions

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Saldana, PhD, Principal Investigator — Chestnut Health Systems
Locations (1):
- Chestnut Health Systems, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of the HEAL Initiative, this study will follow the data sharing protocol set up by the Collaborating Center. Plan development currently in process.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2022 will be the first data upload. This will occur annually until study completion. Data will be available to the HEAL collaborative indefinitely.
Access Criteria: Must be a member of the NIDA HEAL Prevention Collaborative.

DOCUMENTS (1):
  • Informed Consent Form (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT05380440/ICF_000.pdf